CLINICAL TRIAL: NCT02082080
Title: Prevention and Control of Obesity in Primary School Children in Tehran
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: adjazayery
Record Dates: First submitted 2013-12-27; First posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Childhood Obesity Prevention
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obese and overweight children, education (Active Comparator): Overweight and obese school children in grades 5 and 6
  Interventions: Other: Education; Other: Social support
- Obese and overweight children (No Intervention)

INTERVENTIONS:
Other: Education
  Arms: Obese and overweight children, education
Other: Social support
  Arms: Obese and overweight children, education

SUMMARY:
This study evaluates the effect of an interventional model for preventing and controlling overweight and obesity in male and female fifth-graders. First, based on WHO (World Health Organization) references obese (BMI-Z score ≥ 2) and overweight (BMI-Z score ≥ 1) students from 12 primary schools (randomly allocated to 6 intervention and 6 comparison) will be screened. Then from the screened students 30 students with the following inclusion criteria will be recruited: not metabolically ill, not on a weight losing diet and not professionally athlete. For selected students BMI-Z score as primary outcome will be calculated. Demographic data, as well as data on waist and hip circumference, triceps skin-fold thickness, food intake for 3 days (2 ordinary week days and 1 weekend) and physical activity will be collected at the beginning and at end of the 6-month intervention. The approach of the study will be Health Promoting Schools. The intervention includes three components, i.e., nutrition education (students and parents), increased physical activity, and changing environment (food items offered in schools' canteens). Nutrition education will be imparted (a 30-minute session per week) by health instructors; physical activity will be done under the supervision of the school coaches (2 one-hour sessions per week). Parents' education (a 1.5-hour session) will be monthly. Finally the efficacy of the intervention will be determined and reported.

ELIGIBILITY:
Inclusion Criteria:

* BMI-Z-Score> or =1 (WHO)
* Students in the fifth or sixth grades

Exclusion Criteria:

* Metabolic disorders (hypo or hyperthyroidism)
* Any disease which interfere with adherence to the intervention
* Intake of any appetite-reducing drug
* Doing professional sports
* Being on a weight reduction diet

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on the 11-point Short Pain Scale (SPS-11) at week 24 Change from baseline BMI (Body Mass Index) at 6 months | Baseline, month 6

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran